CLINICAL TRIAL: NCT02843997
Title: Endophenotype Characterization of a Family Psychiatric Disorder of the Bipolar Spectrum, With an Autosomal Dominant Expression
Brief Title: Endophenotype Characterization of a Family Psychiatric Disorder
Acronym: EnBiGen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC14.321
Record Dates: First submitted 2016-07-11; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer
Keywords: Bipolar disorder; Endophenotype; Family; Autosomal dominant expression; Sequencing; Heritability
MeSH Terms: conditions — Bipolar Disorder | interventions — Endophenotypes; Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other): Members of a family
  Interventions: Genetic: Endophenotype and sequencing

INTERVENTIONS:
Genetic: Endophenotype and sequencing — Draw an endophenotype and genetic study

SUMMARY:
Bipolar disorder is a chronic and frequent mood pathology, that impacts on emotional and socio-professional life of sick subjects, and also increase mortality by suicide. Suicide is considered as a bipolar disorder result.

The main goal of this study is the endophenotype characterization from a clinical and cognitive point of view, of a bipolar spectrum's disorder present in a family, and then highlight a mutation of one of the genes involved is this disorder.

DETAILED DESCRIPTION:
Heritability of bipolar disorder is now well established, but seems to be multifactorial in most of the cases.

The use of an endophenotype characterized in a family presenting numerous bipolar sufferers enable to reflect the expression of simpler genetic variants than those involved in the disease, and might enable the identification of genes involved in the etiopathogenesis of this endophenotype.

ELIGIBILITY:
Inclusion Criteria:

* Members of a family adult (more than 18 years)
* Signed informed consents
* Registered to a French social security or possesor of the European Health Insurance Card

Exclusion Criteria:

Clinical part :

* Refusal to sign the participation study consent.
* Organic affection likely to affect cognitive abilities and brain structures or acute decompensation of a bipolar disorder.

Genetic part :

* Refusal to sign the genetic sample consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological evaluations tests | One day
  Neuropsychological evaluations (about one hour) :
  TMT (Trail Making Test) A and B, Stroop VFT (Visual Field Testing), DST (Dyslexia Screening Test) Tower of London test Hayling, CPT (continuous performance task) CVLT (California Verbal Learning Test) tests.
Eye tracking. | One hour
  The volunteer will follow an instruction according to the color seen on a screen.
  This instruction is to look at the side where there is a flashlight and to look at the opopsite if the light is unbroken.
  Mistakes will be count.
Blood sampling | 3 minutes
  Genetic sample for extraction of DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Holtzmann, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Adida M, Azorin JM, Fakra E, Belzeaux R, Kaladjian A, Pomietto P, Correard N. [Schizophrenia and/or bipolar disorder: neurobiological endophenotypes]. Encephale. 2012 Dec;38 Suppl 3:S98-102. doi: 10.1016/S0013-7006(12)70086-6. French. PMID 23279996
- [Background] Ancin I, Santos JL, Teijeira C, Sanchez-Morla EM, Bescos MJ, Argudo I, Torrijos S, Vazquez-Alvarez B, De La Vega I, Lopez-Ibor JJ, Barabash A, Cabranes-Diaz JA. Sustained attention as a potential endophenotype for bipolar disorder. Acta Psychiatr Scand. 2010 Sep;122(3):235-45. doi: 10.1111/j.1600-0447.2009.01532.x. Epub 2010 Jan 25. PMID 20105148
- [Background] Badner JA, Koller D, Foroud T, Edenberg H, Nurnberger JI Jr, Zandi PP, Willour VL, McMahon FJ, Potash JB, Hamshere M, Grozeva D, Green E, Kirov G, Jones I, Jones L, Craddock N, Morris D, Segurado R, Gill M, Sadovnick D, Remick R, Keck P, Kelsoe J, Ayub M, MacLean A, Blackwood D, Liu CY, Gershon ES, McMahon W, Lyon GJ, Robinson R, Ross J, Byerley W. Genome-wide linkage analysis of 972 bipolar pedigrees using single-nucleotide polymorphisms. Mol Psychiatry. 2012 Jul;17(8):818-26. doi: 10.1038/mp.2011.89. Epub 2011 Jul 19. PMID 21769101
- [Background] Bertelsen A, Harvald B, Hauge M. A Danish twin study of manic-depressive disorders. Br J Psychiatry. 1977 Apr;130:330-51. doi: 10.1192/bjp.130.4.330. PMID 558030
- [Background] Beynel L, Chauvin A, Guyader N, Harquel S, Szekely D, Bougerol T, Marendaz C. What saccadic eye movements tell us about TMS-induced neuromodulation of the DLPFC and mood changes: a pilot study in bipolar disorders. Front Integr Neurosci. 2014 Aug 19;8:65. doi: 10.3389/fnint.2014.00065. eCollection 2014. PMID 25191234
- [Background] Billieux J, Rochat L, Ceschi G, Carre A, Offerlin-Meyer I, Defeldre AC, Khazaal Y, Besche-Richard C, Van der Linden M. Validation of a short French version of the UPPS-P Impulsive Behavior Scale. Compr Psychiatry. 2012 Jul;53(5):609-15. doi: 10.1016/j.comppsych.2011.09.001. Epub 2011 Oct 27. PMID 22036009
- [Background] Brent D. In search of endophenotypes for suicidal behavior. Am J Psychiatry. 2009 Oct;166(10):1087-9. doi: 10.1176/appi.ajp.2009.09081131. No abstract available. PMID 19797437
- [Background] Cardno AG, Marshall EJ, Coid B, Macdonald AM, Ribchester TR, Davies NJ, Venturi P, Jones LA, Lewis SW, Sham PC, Gottesman II, Farmer AE, McGuffin P, Reveley AM, Murray RM. Heritability estimates for psychotic disorders: the Maudsley twin psychosis series. Arch Gen Psychiatry. 1999 Feb;56(2):162-8. doi: 10.1001/archpsyc.56.2.162. PMID 10025441
- [Background] Cermolacce M, Fakra E, Belzeaux R, Adida M, Azorin JM. [Schizophrenic and bipolar endophenotypes: the clinician's point of view]. Encephale. 2012 Dec;38 Suppl 3:S57-61. doi: 10.1016/S0013-7006(12)70078-7. French. PMID 23279988
- [Background] Chauvin, A. et al. Saccadic inhibition - A trait biomarker of bipolar disorder. 16th Annual conference of the International Society for Bipolar Disorder (2014).
- [Background] Chiaroni P, Hantouche EG, Gouvernet J, Azorin JM, Akiskal HS. The cyclothymic temperament in healthy controls and familially at risk individuals for mood disorder: endophenotype for genetic studies? J Affect Disord. 2005 Mar;85(1-2):135-45. doi: 10.1016/j.jad.2003.12.010. PMID 15780684
- [Background] Courtet P, Gottesman II, Jollant F, Gould TD. The neuroscience of suicidal behaviors: what can we expect from endophenotype strategies? Transl Psychiatry. 2011;1(5):e7-. doi: 10.1038/tp.2011.6. PMID 21761009
- [Background] Daban C, Mathieu F, Raust A, Cochet B, Scott J, Etain B, Leboyer M, Bellivier F. Is processing speed a valid cognitive endophenotype for bipolar disorder? J Affect Disord. 2012 Jun;139(1):98-101. doi: 10.1016/j.jad.2012.02.028. Epub 2012 Mar 18. PMID 22429444
- [Background] Drancourt N, Etain B, Lajnef M, Henry C, Raust A, Cochet B, Mathieu F, Gard S, Mbailara K, Zanouy L, Kahn JP, Cohen RF, Wajsbrot-Elgrabli O, Leboyer M, Scott J, Bellivier F. Duration of untreated bipolar disorder: missed opportunities on the long road to optimal treatment. Acta Psychiatr Scand. 2013 Feb;127(2):136-44. doi: 10.1111/j.1600-0447.2012.01917.x. Epub 2012 Aug 20. PMID 22901015
- [Background] Duffy A, Lewitzka U, Doucette S, Andreazza A, Grof P. Biological indicators of illness risk in offspring of bipolar parents: targeting the hypothalamic-pituitary-adrenal axis and immune system. Early Interv Psychiatry. 2012 May;6(2):128-37. doi: 10.1111/j.1751-7893.2011.00323.x. Epub 2011 Dec 20. PMID 22182213
- [Background] Edvardsen J, Torgersen S, Roysamb E, Lygren S, Skre I, Onstad S, Oien PA. Heritability of bipolar spectrum disorders. Unity or heterogeneity? J Affect Disord. 2008 Mar;106(3):229-40. doi: 10.1016/j.jad.2007.07.001. Epub 2007 Aug 9. PMID 17692389
- [Background] Ferrari AJ, Norman RE, Freedman G, Baxter AJ, Pirkis JE, Harris MG, Page A, Carnahan E, Degenhardt L, Vos T, Whiteford HA. The burden attributable to mental and substance use disorders as risk factors for suicide: findings from the Global Burden of Disease Study 2010. PLoS One. 2014 Apr 2;9(4):e91936. doi: 10.1371/journal.pone.0091936. eCollection 2014. PMID 24694747
- [Background] Ferreira MA, O'Donovan MC, Meng YA, Jones IR, Ruderfer DM, Jones L, Fan J, Kirov G, Perlis RH, Green EK, Smoller JW, Grozeva D, Stone J, Nikolov I, Chambert K, Hamshere ML, Nimgaonkar VL, Moskvina V, Thase ME, Caesar S, Sachs GS, Franklin J, Gordon-Smith K, Ardlie KG, Gabriel SB, Fraser C, Blumenstiel B, Defelice M, Breen G, Gill M, Morris DW, Elkin A, Muir WJ, McGhee KA, Williamson R, MacIntyre DJ, MacLean AW, St CD, Robinson M, Van Beck M, Pereira AC, Kandaswamy R, McQuillin A, Collier DA, Bass NJ, Young AH, Lawrence J, Ferrier IN, Anjorin A, Farmer A, Curtis D, Scolnick EM, McGuffin P, Daly MJ, Corvin AP, Holmans PA, Blackwood DH, Gurling HM, Owen MJ, Purcell SM, Sklar P, Craddock N; Wellcome Trust Case Control Consortium. Collaborative genome-wide association analysis supports a role for ANK3 and CACNA1C in bipolar disorder. Nat Genet. 2008 Sep;40(9):1056-8. doi: 10.1038/ng.209. PMID 18711365
- [Background] Frey BN, Andreazza AC, Houenou J, Jamain S, Goldstein BI, Frye MA, Leboyer M, Berk M, Malhi GS, Lopez-Jaramillo C, Taylor VH, Dodd S, Frangou S, Hall GB, Fernandes BS, Kauer-Sant'Anna M, Yatham LN, Kapczinski F, Young LT. Biomarkers in bipolar disorder: a positional paper from the International Society for Bipolar Disorders Biomarkers Task Force. Aust N Z J Psychiatry. 2013 Apr;47(4):321-32. doi: 10.1177/0004867413478217. Epub 2013 Feb 14. PMID 23411094
- [Background] Geoffroy PA, Etain B, Jamain S, Bellivier F, Leboyer M. [Early onset bipolar disorder: validation from admixture analyses and biomarkers]. Can J Psychiatry. 2013 Apr;58(4):240-8. doi: 10.1177/070674371305800410. French. PMID 23547648
- [Background] Glahn DC, Almasy L, Barguil M, Hare E, Peralta JM, Kent JW Jr, Dassori A, Contreras J, Pacheco A, Lanzagorta N, Nicolini H, Raventos H, Escamilla MA. Neurocognitive endophenotypes for bipolar disorder identified in multiplex multigenerational families. Arch Gen Psychiatry. 2010 Feb;67(2):168-77. doi: 10.1001/archgenpsychiatry.2009.184. PMID 20124116
- [Background] Gooding DC, Basso MA. The tell-tale tasks: a review of saccadic research in psychiatric patient populations. Brain Cogn. 2008 Dec;68(3):371-90. doi: 10.1016/j.bandc.2008.08.024. Epub 2008 Oct 23. PMID 18950927
- [Background] Gottesman II, Gould TD. The endophenotype concept in psychiatry: etymology and strategic intentions. Am J Psychiatry. 2003 Apr;160(4):636-45. doi: 10.1176/appi.ajp.160.4.636. PMID 12668349
- [Background] Harvey AG. Sleep and circadian rhythms in bipolar disorder: seeking synchrony, harmony, and regulation. Am J Psychiatry. 2008 Jul;165(7):820-9. doi: 10.1176/appi.ajp.2008.08010098. Epub 2008 Jun 2. PMID 18519522
- [Background] Hasler G, Drevets WC, Gould TD, Gottesman II, Manji HK. Toward constructing an endophenotype strategy for bipolar disorders. Biol Psychiatry. 2006 Jul 15;60(2):93-105. doi: 10.1016/j.biopsych.2005.11.006. Epub 2006 Jan 9. PMID 16406007
- [Background] Houenou J, Frommberger J, Carde S, Glasbrenner M, Diener C, Leboyer M, Wessa M. Neuroimaging-based markers of bipolar disorder: evidence from two meta-analyses. J Affect Disord. 2011 Aug;132(3):344-55. doi: 10.1016/j.jad.2011.03.016. Epub 2011 Apr 5. PMID 21470688
- [Background] Hranov LG, Marinova P, Stoyanova M, Pandova M, Hranov G. Bipolar disorder - from endophenotypes to treatment. Psychiatr Danub. 2013 Sep;25(3):284-91. PMID 24048399
- [Background] Jimenez-Trevino L, Blasco-Fontecilla H, Braquehais MD, Ceverino-Dominguez A, Baca-Garcia E. Endophenotypes and suicide behaviour. Actas Esp Psiquiatr. 2011 Jan-Feb;39(1):61-9. Epub 2011 Jan 1. PMID 21274823
- [Background] Jollant F, Guillaume S, Jaussent I, Bellivier F, Leboyer M, Castelnau D, Malafosse A, Courtet P. Psychiatric diagnoses and personality traits associated with disadvantageous decision-making. Eur Psychiatry. 2007 Oct;22(7):455-61. doi: 10.1016/j.eurpsy.2007.06.001. Epub 2007 Aug 30. PMID 17764910
- [Background] Judd LL, Schettler PJ, Akiskal HS, Maser J, Coryell W, Solomon D, Endicott J, Keller M. Long-term symptomatic status of bipolar I vs. bipolar II disorders. Int J Neuropsychopharmacol. 2003 Jun;6(2):127-37. doi: 10.1017/S1461145703003341. PMID 12890306
- [Background] Kendler KS. Twin studies of psychiatric illness. Current status and future directions. Arch Gen Psychiatry. 1993 Nov;50(11):905-15. doi: 10.1001/archpsyc.1993.01820230075007. No abstract available. PMID 8215816
- [Background] Kendler KS. Twin studies of psychiatric illness: an update. Arch Gen Psychiatry. 2001 Nov;58(11):1005-14. doi: 10.1001/archpsyc.58.11.1005. PMID 11695946
- [Background] Latalova K, Prasko J, Diveky T, Velartova H. Cognitive impairment in bipolar disorder. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2011 Mar;155(1):19-26. doi: 10.5507/bp.155.2011.003. PMID 21475373
- [Background] Lombardo LE, Bearden CE, Barrett J, Brumbaugh MS, Pittman B, Frangou S, Glahn DC. Trait impulsivity as an endophenotype for bipolar I disorder. Bipolar Disord. 2012 Aug;14(5):565-70. doi: 10.1111/j.1399-5618.2012.01035.x. Epub 2012 Jul 16. PMID 22805501
- [Background] Mahon K, Perez-Rodriguez MM, Gunawardane N, Burdick KE. Dimensional endophenotypes in bipolar disorder: affective dysregulation and psychosis proneness. J Affect Disord. 2013 Nov;151(2):695-701. doi: 10.1016/j.jad.2013.08.003. Epub 2013 Aug 14. PMID 23993441
- [Background] Malsert J, Guyader N, Chauvin A, Polosan M, Poulet E, Szekely D, Bougerol T, Marendaz C. Antisaccades as a follow-up tool in major depressive disorder therapies: a pilot study. Psychiatry Res. 2012 Dec 30;200(2-3):1051-3. doi: 10.1016/j.psychres.2012.05.007. Epub 2012 May 28. PMID 22648007
- [Background] Malsert J, Guyader N, Chauvin A, Polosan M, Szekely D, Bougerol T, Marendaz C. Saccadic performance and cortical excitability as trait-markers and state-markers in rapid cycling bipolar disorder: a two-case follow-up study. Front Psychiatry. 2013 Jan 4;3:112. doi: 10.3389/fpsyt.2012.00112. eCollection 2012. PMID 23293609
- [Background] Mann JJ, Arango VA, Avenevoli S, Brent DA, Champagne FA, Clayton P, Currier D, Dougherty DM, Haghighi F, Hodge SE, Kleinman J, Lehner T, McMahon F, Moscicki EK, Oquendo MA, Pandey GN, Pearson J, Stanley B, Terwilliger J, Wenzel A. Candidate endophenotypes for genetic studies of suicidal behavior. Biol Psychiatry. 2009 Apr 1;65(7):556-63. doi: 10.1016/j.biopsych.2008.11.021. Epub 2009 Feb 7. PMID 19201395
- [Background] Marian AJ. Sequencing your genome: what does it mean? Methodist Debakey Cardiovasc J. 2014 Jan-Mar;10(1):3-6. doi: 10.14797/mdcj-10-1-3. PMID 24932355
- [Background] Mazzola-Pomietto P, Azorin JM, Belzeaux R, Fakra E, Adida M, Kaladjian A. [Are variations of structural neuro-anatomy promising endophenotype candidates in bipolar disorder?]. Encephale. 2012 Dec;38 Suppl 3:S75-80. doi: 10.1016/S0013-7006(12)70082-9. French. PMID 23279992
- [Background] McGirr A, Alda M, Seguin M, Cabot S, Lesage A, Turecki G. Familial aggregation of suicide explained by cluster B traits: a three-group family study of suicide controlling for major depressive disorder. Am J Psychiatry. 2009 Oct;166(10):1124-34. doi: 10.1176/appi.ajp.2009.08111744. Epub 2009 Sep 15. PMID 19755577
- [Background] Mendlowicz MV, Jean-Louis G, Kelsoe JR, Akiskal HS. A comparison of recovered bipolar patients, healthy relatives of bipolar probands, and normal controls using the short TEMPS-A. J Affect Disord. 2005 Mar;85(1-2):147-51. doi: 10.1016/j.jad.2004.01.012. PMID 15780685
- [Background] Merikangas KR, Akiskal HS, Angst J, Greenberg PE, Hirschfeld RM, Petukhova M, Kessler RC. Lifetime and 12-month prevalence of bipolar spectrum disorder in the National Comorbidity Survey replication. Arch Gen Psychiatry. 2007 May;64(5):543-52. doi: 10.1001/archpsyc.64.5.543. PMID 17485606
- [Background] Mortensen PB, Pedersen CB, Melbye M, Mors O, Ewald H. Individual and familial risk factors for bipolar affective disorders in Denmark. Arch Gen Psychiatry. 2003 Dec;60(12):1209-15. doi: 10.1001/archpsyc.60.12.1209. PMID 14662553
- [Background] Myles-Worsley M, Tiobech J, Browning SR, Korn J, Goodman S, Gentile K, Melhem N, Byerley W, Faraone SV, Middleton FA. Deletion at the SLC1A1 glutamate transporter gene co-segregates with schizophrenia and bipolar schizoaffective disorder in a 5-generation family. Am J Med Genet B Neuropsychiatr Genet. 2013 Mar;162B(2):87-95. doi: 10.1002/ajmg.b.32125. Epub 2013 Jan 22. PMID 23341099
- [Background] Parmentier C, Etain B, Yon L, Misson H, Mathieu F, Lajnef M, Cochet B, Raust A, Kahn JP, Wajsbrot-Elgrabli O, Cohen R, Henry C, Leboyer M, Bellivier F. Clinical and dimensional characteristics of euthymic bipolar patients with or without suicidal behavior. Eur Psychiatry. 2012 Nov;27(8):570-6. doi: 10.1016/j.eurpsy.2011.05.005. Epub 2011 Oct 5. PMID 21978427
- [Background] Peters E, Joseph S, Day S, Garety P. Measuring delusional ideation: the 21-item Peters et al. Delusions Inventory (PDI). Schizophr Bull. 2004;30(4):1005-22. doi: 10.1093/oxfordjournals.schbul.a007116. PMID 15954204
- [Background] Ross J, Berrettini W, Coryell W, Gershon ES, Badner JA, Kelsoe JR, McInnis MG, McMahon FJ, Murphy DL, Nurnberger JI Jr, Foroud T, Rice JP, Scheftner WB, Zandi P, Edenberg H, Byerley W. Genome-wide parametric linkage analyses of 644 bipolar pedigrees suggest susceptibility loci at chromosomes 16 and 20. Psychiatr Genet. 2008 Aug;18(4):191-8. doi: 10.1097/YPG.0b013e3283050aa5. PMID 18628681
- [Background] Schurhoff F, Szoke A, Meary A, Bellivier F, Rouillon F, Pauls D, Leboyer M. Familial aggregation of delusional proneness in schizophrenia and bipolar pedigrees. Am J Psychiatry. 2003 Jul;160(7):1313-9. doi: 10.1176/appi.ajp.160.7.1313. PMID 12832247
- [Background] Smoller JW, Finn CT. Family, twin, and adoption studies of bipolar disorder. Am J Med Genet C Semin Med Genet. 2003 Nov 15;123C(1):48-58. doi: 10.1002/ajmg.c.20013. PMID 14601036
- [Background] St Clair D, Blackwood D, Muir W, Carothers A, Walker M, Spowart G, Gosden C, Evans HJ. Association within a family of a balanced autosomal translocation with major mental illness. Lancet. 1990 Jul 7;336(8706):13-6. doi: 10.1016/0140-6736(90)91520-k. PMID 1973210
- [Background] Vazquez GH, Kahn C, Schiavo CE, Goldchluk A, Herbst L, Piccione M, Saidman N, Ruggeri H, Silva A, Leal J, Bonetto GG, Zaratiegui R, Padilla E, Vilaprino JJ, Calvo M, Guerrero G, Strejilevich SA, Cetkovich-Bakmas MG, Akiskal KK, Akiskal HS. Bipolar disorders and affective temperaments: a national family study testing the "endophenotype" and "subaffective" theses using the TEMPS-A Buenos Aires. J Affect Disord. 2008 May;108(1-2):25-32. doi: 10.1016/j.jad.2007.09.011. Epub 2007 Nov 19. PMID 18006072
- [Background] Verdoux H, van Os J, Maurice-Tison S, Gay B, Salamon R, Bourgeois M. Is early adulthood a critical developmental stage for psychosis proneness? A survey of delusional ideation in normal subjects. Schizophr Res. 1998 Feb 9;29(3):247-54. doi: 10.1016/s0920-9964(97)00095-9. PMID 9516665
- [Background] WHO. The world health report 2001.
- [Background] Xu G, Lu W, Ouyang H, Dang Y, Guo Y, Miao G, Bessonov D, Akiskal KK, Akiskal HS, Lin K. Association of affective temperaments measured by TEMPS-a with cognitive deficits in patients with bipolar disorder. J Affect Disord. 2014 Jun;161:109-15. doi: 10.1016/j.jad.2014.03.005. Epub 2014 Mar 21. PMID 24751317